CLINICAL TRIAL: NCT04792762
Title: Physiology of GIP(1-30)NH2 in Humans
Acronym: GA-11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-17039726
Record Dates: First submitted 2021-03-06; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — gastric inhibitory polypeptide (1-42); Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GIP(1-42) (Experimental)
  Interventions: Other: GIP(1-42)
- GIP(1-30)NH2 (Experimental)
  Interventions: Other: GIP(1-30)NH2
- Placebo (Placebo Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Other: GIP(1-30)NH2 — Intravenous administration of the peptide hormone GIP(1-30)NH2 during a stepwise glucose clamp
  Arms: GIP(1-30)NH2
Other: GIP(1-42) — Intravenous administration of the peptide hormone GIP(1-42) during a stepwise glucose clamp
  Arms: GIP(1-42)
Other: Saline — Intravenous administration of saline during a stepwise glucose clamp
  Arms: Placebo

SUMMARY:
Glucose-dependent insulinotropic polypeptide (GIP) is a gut-derived incretin hormone that affects glucose, lipid and bone metabolism. Secretion of GIP into the blood stream from enteroendocrine cells is stimulated bu nutrients in the gut lumen and results in potentiation of glucose stimulated insulin secretion from the pancreas. The objective of this study is to investigate the physiology of GIP(1-30)NH2 in humans with insulin secretion as the primary endpoint. Furthermore the effects on on plasma/serum levels of glucagon, C-peptide, glucose, bone markers (CTX and P1NP) will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men of Northern European descent
* BMI: 19-25 kg/m2
* Stable body weight (±5%) in the last three months

Exclusion Criteria:

* Treatment with medication or dietary supplements that cannot be paused for 12 hours
* More than 14 units of alcohol per week or abuse of narcotics
* Established liver disease and/or plasma alanine aminotransferase (ALT) ≥3 × normal value and/or INR outside the normal range
* Renal impairment (eGFR <60 ml/min/1.73 m2)
* Severe arteriosclerotic heart disease or severe heart failure (NYHA group III or IV)
* Low blood count (haemoglobin <8.3 mol/l)
* Special diet or planned body weight change before the trial period
* First-degree relatives with diabetes
* Participation in other clinical experiments with medication
* Any disease/condition that the investigators estimate disturbing for the participation in the experiment

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2019-06-09 (Actual)

PRIMARY OUTCOMES:
Insulin | Up to 3 months

SECONDARY OUTCOMES:
Glucagon | Up to 3 months
C-peptide | Up to 3 months
Glucose | Up to 3 months
CTX | Up to 3 months
P1NP | Up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Metabolic Physiology, Hellerup, Denmark